CLINICAL TRIAL: NCT04672057
Title: Investigation of the Spatio-temporal Gait Parameters in Individuals With Hemiparesis: Effect of Lateralization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gulsum Tikac, Principal Investigator, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Gait Parameter In Hemiparetics
Record Dates: First submitted 2020-12-06; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hemiparesis
Keywords: Hemiparesis; Lateralization; Spatio-temporal analysis; Gait
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Right hemiparetics (Active Comparator): right-sided affected hemiparetic individuals
  Interventions: Other: assessment of gait parameters
- Left hemiparetics (Active Comparator): left-sided affected hemiparetic individuals
  Interventions: Other: assessment of gait parameters
- Control (Active Comparator): healthy individuals
  Interventions: Other: assessment of gait parameters

INTERVENTIONS:
Other: assessment of gait parameters — Gait parameters have been recourded with the use of BTS G-Walk Wireless Digital Walking Analysis System on a 10-meter smooth walking area.

SUMMARY:
The aim of this study was to investigate the effect of lateralization on the spatio-temporal characteristics of gait in individuals with hemiparesis.

DETAILED DESCRIPTION:
A total of 108 individuals within the age range of 20-65 and 36 of whom are right hemiparetic (Group1; 16F, 20M), 36 of whom are left hemiparetic (Group2; 16F, 20M) and 36 of whom are healthy (Group3; 19F, 17M) have been included in the study. BTS G-Walk Gait Analysis System has been used to assess the spatio-temporal gait characteristics.

ELIGIBILITY:
Inclusion Criteria:

for the hemiparetic individuals

* Being between the ages of 20-65,
* Having a stroke for the first time and one-sidedly,
* Having a stable clinical state,
* Having no cognitive disorder (Hodkinson Mental Test ≥ 8),
* Having ≤ 3 from Modified Rankin Score,
* Having no problems with vision and hearing.

for the healthy control group;

* Being between the ages of 20-65
* Having no neurological, musculosceletal, cardiac and cognitive problems that was undergone before and may affect walking.

Exclusion Criteria:

* The existence of vision and hearing problems in both study and control groups,
* The existence of orthopedic, neurological and psychiatric problems that may affect walking.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-07-08 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
assessment of gait between in right and left hemiparetics | Measurement time is 10 minutes. Only one measurement was made.
  A port was attached to the patient's L5-S1 level. In the gait analysis system, the results was transferred to the computer via bluetooth with the analysis port. The resulting report was generated automatically. The report measured gait speed, cadence, right and left step length, right and left stride length, double and single stride length, pelvic rotation, pelvic tilt, and pelvic oblique.

SECONDARY OUTCOMES:
assessment of gait between in hemiparetic and healthy individuals | Measurement time is 10 minutes. Only one measurement was made.
  A port was attached to the patient's L5-S1 level. In the gait analysis system, the results was transferred to the computer via bluetooth with the analysis port. The resulting report was generated automatically. The report measured gait speed, cadence, right and left step length, right and left stride length, double and single stride length, pelvic rotation, pelvic tilt, and pelvic oblique.

CONTACTS AND LOCATIONS:
Overall Officials: Gulsum Tikac, MSc Pt, Principal Investigator — Pamukkale University; Filiz Altuğ, Prof Dr, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No